CLINICAL TRIAL: NCT03354104
Title: Tunnel Technique With Emdogain® in Addition to Connective Tissue Graft Compared With Connective Tissue Graft Alone for the Treatment of Gingival (Periodontal?) Recessions: a Randomized Clinical Trial.
Brief Title: Tunnel Technique With Emdogain® in Addition to Connective Tissue Graft Compared With Connective Tissue Graft Alone for the Treatment of Gingival Recessions: a Randomized Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WUM.PERIO.01
Record Dates: First submitted 2017-11-08; First posted 2017-11-27 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recession coverage with connective tissue graft + Emdogain® (Experimental): A modified microsurgical tunnel technique by Zuhr et al. (2007). Initial sulcular incisions with a microsurgical blade are followed by a split-thickness buccal flap preparations using the tunneling knives. The preparation is extended into the mucosal tissue to gain sufficient flap mobility. The papillary regions are detached in their buccal aspects with the periosteum. The root surfaces are applied with 24% EDTA (PrefGel®, Straumann, Basel, Switzerland) for 2 minutes and then washed with saline. Subsequently, EMD (Emdogain®, Straumann, Basel, Switzerland) is applied on root surfaces. The graft is inserted into the tunnel and stabilized with absorbable suspensory sutures. The buccal flap is advanced coronally and stabilized with non-absorbable suspensory sutures.
  Interventions: Device: The tunnel technique for root coverage with Emdogain
- Recession coverage with connective tissue graft (Active Comparator): Procedure: A modified microsurgical tunnel technique by Zuhr et al. (2007). Initial sulcular incisions with a microsurgical blade are followed by a split-thickness buccal flap preparations using the tunneling knives. The preparation is extended into the mucosal tissue to gain sufficient flap mobility. The papillary regions are detached in their buccal aspects with the periosteum. The graft is inserted into the tunnel and stabilized with absorbable suspensory sutures. The buccal flap is advanced coronally and stabilized with non-absorbable suspensory sutures.
  Interventions: Device: The tunnel technique for root coverage without Emdogain

INTERVENTIONS:
Device: The tunnel technique for root coverage with Emdogain — The tunnel technique for root coverage with Emdogain
  Arms: Recession coverage with connective tissue graft + Emdogain®
Device: The tunnel technique for root coverage without Emdogain — The tunnel technique for root coverage without Emdogain
  Arms: Recession coverage with connective tissue graft

SUMMARY:
Microsurgical tunneling flap procedures using connective tissue grafts (CTG) are predictable for treating teeth with gingival recessions. Enamel matrix derivatives (EMD) can be used as an alternative to the aforementioned gold standard. The aim of this study is to evaluate clinically the use of tunnel technique with EMD applied group in addition to CTG and the same technique with CTG group for the treatment of multiple gingival recessions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Bilateral multiple gingival recessions in homologous teeth

Exclusion Criteria:

* Full-mouth plaque index ≥ 20% (Ainamo & Bay 1975)
* Full-mouth sulcus bleeding index ≥ 15% (Mühlemann & Son 1971)
* Smoking
* Systemic diseases with compromised healing potential of infectious diseases
* Drugs affecting periodontal health / healing
* Pregnant and lactating females
* Previous periodontal surgery in the area

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-01-05 (Estimated); Study Completion 2019-05-05 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) | 6 months after surgery
  Distance from the cementoenamel junction to the bottom of the gingival sulcus

SECONDARY OUTCOMES:
Recession height (RH) | 6 months after surgery
  Distance from the cementoenamel junction to the gingival margin
Recession width (RW) | 6 months after surgery
  Distance measured horizontally at cementoenamel junction level from one border of the recession to another
Width of keratinized tissue (WKT) | 6 months after surgery
  Distance between the most apical point of the gingival margin and the mucogingival junction
Thickness of keratinized tissue (TKT) | 6 months after surgery
  Thickness of the gingiva measured 2 mm apical to the gingival margin
Average recession coverage (ARC) | 6 months after surgery
  The percentage of covered recession area
Complete recession coverage | 6 months after surgery
  The percentage of sites with complete root coverage

OTHER OUTCOMES:
Probing pocket depth (PPD) | 6 months after surgery
  Distance from the gingival margin to the bottom of the gingival sulcus
Root coverage esthetic score (RES) | 6 months after surgery
  A score including root coverage, marginal gingival tissue contour, mucogingival junction alignment, soft tissue texture and gingival colour according to Cairo et al. (1999)
Post surgical pain and swelling | 1, 2, 4, 7 and 14 days after surgery
  Questionnaire about post surgical pain and swelling using a Visual Analog Scale with values 0 (no pain / swelling), 1, 2, 3, 4, 5(moderate pain/swelling), 6, 7, 8, 9, 10 (worst pain / swelling). Lower values represent lower post surgical discomfort and are considered better.
Patient's satisfaction with treatment | 6 months after surgery
  Questionnaire about patient's esthetic perception of gingiva and overall satisfaction using a Visual Analog Scale from 0 (dissatisfaction with esthetic outcome), 2, 3, 4, 5 (moderate satisfaction with easthetic outcome), 6, 7, 8, 9, 10 (best satisfaction with esthetic outcome). Higher values are considered better.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology and Oral Mucosa Diseases, Medical University of Warsaw, Warsaw, Mazowsze, Poland

REFERENCES:
- [Derived] Gorski B, Szerszen M, Kaczynski T. Effect of 24% EDTA root conditioning on the outcome of modified coronally advanced tunnel technique with subepithelial connective tissue graft for the treatment of multiple gingival recessions: a randomized clinical trial. Clin Oral Investig. 2022 Feb;26(2):1761-1772. doi: 10.1007/s00784-021-04151-9. Epub 2021 Aug 24. PMID 34431001